CLINICAL TRIAL: NCT01613911
Title: A Combined fMRI and Electrophysiological Study of Human Sensory Perception
Brief Title: Study of Human Sensory Perception
Status: Completed | Type: Observational
Sponsor: Swedish Medical Center (Other)
Collaborators: Weizmann Institute of Science (Other)
Responsible Party: Sponsor
Other Study IDs: 5146S-11
Record Dates: First submitted 2012-06-05; First posted 2012-06-07 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-09

CONDITIONS: Epilepsy
Keywords: Epilepsy; Invasive monitoring; Human sensory perception
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Epileptics having invasive monitoring: People between 10 and 65 years of age with epilepsy and who are coming in to have invasive electrophysiological monitoring.

SUMMARY:
This study will help describe how the human brain works when a person sees something, hears something, learns something, or thinks about something by recording brain activity that occurs when the person does a series of computer tasks. This study will be offered to people who are in the hospital to be monitored for epilepsy by using electrodes placed in the brain. The study will record brain activity that occurs when a patient does a memory task, for example.

DETAILED DESCRIPTION:
Patients who have elected to have invasive electrophysiological monitoring for epileptic activity are invited to participate in this study. While the electrodes are in place, patients are asked to view several scenarios on a laptop computer. During these scenarios, for example, patients are asked to click a mouse button if they see the same picture twice in a row or to remember a film clip of a scooter ride. Trigger points in the computer scenarios are recorded on a separate channel alongside the brain-wave activity to allow correlation between the brain activity and the task requested in the scenario. Using this technique, researchers can determine what areas of the brain were active during recognition or recall activities.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of epilepsy
* Between 10 and 65 years of age
* Scheduled to undergo invasive electrophysiological monitoring as part of a clinical evaluation for epilepsy treatment

Exclusion Criteria:

* None

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People between 10 and 65 years old diagnosed with epilepsy who will have invasive eletrophysioloigcal monitoring as part of a clinical evaluation for epilepsy treatment.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2012-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Reveal induced neuronal activity | Approximately 3 hours over the course of 2-3 days during in-patient invasive electrophysiological monitoring.
  In the preprocessing stage, potential electrical interference will be removed from the raw signal using a linear-phase notch FIR filter. Each electrode will be de-referenced by subtraction of the averaged signal of all the electrodes, thus discarding non-neuronal contributions. Time-frequency decompositions will be calculated for each electrode based on Fourier transform amplitude spectrum in a 160ms sliding window with average step size of 6ms. This process is done per trial and averaged across trials in order to reveal induced neuronal activity, which is not time-locked to the stimuli.

SECONDARY OUTCOMES:
Calculate evoked response potentials. | Approximately 3 hours over the course of 2-3 days during in-patient invasive electrophysiological monitoring.
  Evoked response potentials (ERPs) will be calculated by averaging the raw signal across the presentation of a specific stimulus for each patient, such as all samples of patients watching the movie clip.

CONTACTS AND LOCATIONS:
Locations (1):
- Swedish Medical Center Epilepsy Center, Seattle, Washington, United States

REFERENCES:
- [Background] Allison T, Puce A, Spencer DD, McCarthy G. Electrophysiological studies of human face perception. I: Potentials generated in occipitotemporal cortex by face and non-face stimuli. Cereb Cortex. 1999 Jul-Aug;9(5):415-30. doi: 10.1093/cercor/9.5.415. PMID 10450888
- [Background] Grill-Spector K, Kushnir T, Hendler T, Malach R. The dynamics of object-selective activation correlate with recognition performance in humans. Nat Neurosci. 2000 Aug;3(8):837-43. doi: 10.1038/77754. PMID 10903579
- [Background] Hasson U, Hendler T, Ben Bashat D, Malach R. Vase or face? A neural correlate of shape-selective grouping processes in the human brain. J Cogn Neurosci. 2001 Aug 15;13(6):744-53. doi: 10.1162/08989290152541412. PMID 11564319
- [Background] Hasson U, Nir Y, Levy I, Fuhrmann G, Malach R. Intersubject synchronization of cortical activity during natural vision. Science. 2004 Mar 12;303(5664):1634-40. doi: 10.1126/science.1089506. PMID 15016991
- [Background] Kirsch HE, Sepkuty JP, Crone NE. Multimodal functional mapping of sensorimotor cortex prior to resection of an epileptogenic perirolandic lesion. Epilepsy Behav. 2004 Jun;5(3):407-10. doi: 10.1016/j.yebeh.2004.02.001. PMID 15145312
- [Background] Kleinman JT, Sepkuty JP, Hillis AE, Lenz FA, Heidler-Gary J, Gingis L, Crone NE. Spatial neglect during electrocortical stimulation mapping in the right hemisphere. Epilepsia. 2007 Dec;48(12):2365-8. doi: 10.1111/j.1528-1167.2007.01196.x. Epub 2007 Jul 21. PMID 17645542
- [Background] Kreiman G, Hung CP, Kraskov A, Quiroga RQ, Poggio T, DiCarlo JJ. Object selectivity of local field potentials and spikes in the macaque inferior temporal cortex. Neuron. 2006 Feb 2;49(3):433-45. doi: 10.1016/j.neuron.2005.12.019. PMID 16446146
- [Background] Liu J, Newsome WT. Local field potential in cortical area MT: stimulus tuning and behavioral correlations. J Neurosci. 2006 Jul 26;26(30):7779-90. doi: 10.1523/JNEUROSCI.5052-05.2006. PMID 16870724
- [Background] Logothetis NK. Single units and conscious vision. Philos Trans R Soc Lond B Biol Sci. 1998 Nov 29;353(1377):1801-18. doi: 10.1098/rstb.1998.0333. PMID 9854253
- [Background] Mukamel R, Gelbard H, Arieli A, Hasson U, Fried I, Malach R. Coupling between neuronal firing, field potentials, and FMRI in human auditory cortex. Science. 2005 Aug 5;309(5736):951-4. doi: 10.1126/science.1110913. PMID 16081741
- [Background] Niessing J, Ebisch B, Schmidt KE, Niessing M, Singer W, Galuske RA. Hemodynamic signals correlate tightly with synchronized gamma oscillations. Science. 2005 Aug 5;309(5736):948-51. doi: 10.1126/science.1110948. PMID 16081740
- [Background] Nir Y, Fisch L, Mukamel R, Gelbard-Sagiv H, Arieli A, Fried I, Malach R. Coupling between neuronal firing rate, gamma LFP, and BOLD fMRI is related to interneuronal correlations. Curr Biol. 2007 Aug 7;17(15):1275-85. doi: 10.1016/j.cub.2007.06.066. PMID 17686438
- [Background] Privman E, Nir Y, Kramer U, Kipervasser S, Andelman F, Neufeld MY, Mukamel R, Yeshurun Y, Fried I, Malach R. Enhanced category tuning revealed by intracranial electroencephalograms in high-order human visual areas. J Neurosci. 2007 Jun 6;27(23):6234-42. doi: 10.1523/JNEUROSCI.4627-06.2007. PMID 17553996